CLINICAL TRIAL: NCT00368316
Title: Phase 3 Study (Safety, Immunogenicity and Efficacy) of Improved Shigella Conjugate Vaccines in 1-4 Year Olds in Israel
Brief Title: Safety, Immunogenicity and Efficacy of Shigella Conjugate Vaccines in 1-4 Year Olds in Israel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: The Chaim Sheba Medical Center (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 999900003; OH00-CH-N003 (Registry Identifier: NICHD IRB)
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Shigellosis
Keywords: Dysentery; S. sonnei; Antibody Response; Protection
MeSH Terms: conditions — Dysentery, Bacillary; Dysentery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S. sonnei conjugate vaccine (Experimental): Shigella sonnei O-specific polysaccharide covalently bound to recombinant exoprotein A of Pseudomonas aeruginosa
  Interventions: Biological: Shigella conjugate vaccines
- S. flexneri 2a conjugate vaccine (Experimental): Shigella flexneri 2a O-specific polysaccharide covalently bound to recombinant exoprotein A of pseudomonas aeruginosa
  Interventions: Biological: Shigella conjugate vaccines

INTERVENTIONS:
Biological: Shigella conjugate vaccines — Shigella sonnei-rEPA and Shigella flexneri2a rEPA vaccines
  Other Names: S. sonnei O-SP-rEPA conjugate.; S. flexneri 2a O-SP-rEPA conjugate.

SUMMARY:
Shigellosis remains a serious and frequent disease throughout the world. Development of vaccines has been difficult because shigellae are habitants of and pathogens for humans only and there is no consensus about the mechanism(s) of immunity to this pathogen.

Incomplete, but compelling evidence, indicates that a critical level of serum IgG anti-LPS confers immunity to shigellosis. Important data come from our clinical trial in the Israel Defense Forces (IDF) recruits. A randomized, double-blind, vaccine-controlled study showed that the S. sonnei-rEPA elicited 74% protection against shigellosis occurring about 3 months after vaccination (p=0.001). This vaccine conferred 43% (p=0.04) protection in one company during an outbreak up to 14 days following vaccination suggesting that our Shigella conjugates might be of value in epidemics. The efficacy of S. sonnei-rEPA was correlated with the level of vaccine-induced IgG antibodies.

The highest incidence, morbidity, and mortality of shigellosis is in young children. But serum antibody responsiveness to polysaccharide-based vaccines is age-dependent and infants and young children respond poorly or not at all to both disease and vaccination. The safety and immunogenicity of these Shigella conjugates in 4 to 6 years-old children in Israel was demonstrated. But although the fold rise in anti-LPS was similar in the children, the level of anti-LPS elicited by the conjugates was lower than in adults. We improved the immunogenicity of Shigella conjugates as shown in mice and then in adult humans. Now we apply to evaluate the safety, immunogenicity and efficacy of these improved conjugates in 1 to 4 years-old children in Israel.

In Israel, shigellosis is common especially in children. S. sonnei (Group D) comprise about 60% of the isolates followed by S. flexneri (Group B): Shigella dysenteriae type 1 (Group A) is not found. We propose to administer 2 injections of either S. sonnei-CRM9 or S. flexneri type 2a-rEPAsucc 6 weeks apart in a random double-blind fashion to about 6,000 1 to 4 year-olds. Active surveillance of the vaccinees for enteric infections will be maintained for at least 2 years to evaluate the effect of vaccination.

DETAILED DESCRIPTION:
Shigellosis remains a serious and frequent disease throughout the world. Development of vaccines has been difficult because shigellae are habitants of and pathogens for humans only and there is no consensus about the mechanism/s of immunity to this pathogen.

Incomplete, but compelling evidence, indicates that a critical level of serum IgG anti-LPS confers immunity to shigellosis. A randomized, double-blind, vaccine-controlled study in Israel Defense Force (IDF) recruits showed that the S. sonnei-rEPA elicited 74% protection against shigellosis occurring about 3 months after vaccination (p=0.001). This vaccine also conferred 43% (p=0.04) protection in one company during an outbreak up to 17 days following vaccination suggesting that our Shigella conjugates might be of value in epidemics. The efficacy of S. sonnei-rEPA was correlated with the level of vaccine-induced IgG antibodies.

The highest incidence, morbidity, and mortality of shigellosis is in young children. But serum antibody responsiveness to it is age dependent and infants and young children respond poorly or not at all to polysaccharide antigens following disease, administration of attenuated strains of Shigella or vaccination with whole cell vaccines. The safety and immunogenicity of similar Shigella conjugates in 4 to 7 years-old children in Israel was demonstrated. But, although the fold rise in anti-LPS was similar in the children, the level of anti-LPS elicited by the conjugates was lower than in adults. We improved the immunogenicity of Shigella conjugates as shown in mice and then in adult humans. Now we apply to evaluate the safety, immunogenicity and efficacy of these improved conjugates in 1 to 4 years-old children in Israel. In addition to monitoring the safety and immunogenicity of the two investigational Shigella vaccines, active surveillance of the vaccines for enteric infections wil be maintained for at lest 2 years to evaluate the effect of vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers who are healthy 1-4 year old children whose parents/guardians have read the Information Sheet provided by the Principal Investigator and signed the consent form, and who will be available for follow up.

EXCLUSION CRITERIA: Children with

* chronic diseases receiving medication;
* who have received systemic steroids during the month preceding Shigella vaccination;
* who had severe side effects following vaccinations; and
* those not available for follow up.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2799 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Schneerson, MD, Principal Investigator — PDMI, NICHD, NIH
Locations (2):
- Israel (2):
  - Schneider Childrens Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Tel Aviv

REFERENCES:
- [Background] Development of vaccines against shigellosis: memorandum from a WHO meeting. Bull World Health Organ. 1987;65(1):17-25. PMID 3495364
- [Background] DuPont HL, Hornick RB, Snyder MJ, Libonati JP, Formal SB, Gangarosa EJ. Immunity in shigellosis. II. Protection induced by oral live vaccine or primary infection. J Infect Dis. 1972 Jan;125(1):12-6. doi: 10.1093/infdis/125.1.12. No abstract available. PMID 4550416
- [Background] Taylor DN, Echeverria P, Blaser MJ, Pitarangsi C, Blacklow N, Cross J, Weniger BG. Polymicrobial aetiology of travellers' diarrhoea. Lancet. 1985 Feb 16;1(8425):381-3. doi: 10.1016/s0140-6736(85)91397-2. PMID 2857430
- [Background] Hossain MA, Hasan KZ, Albert MJ. Shigella carriers among non-diarrhoeal children in an endemic area of shigellosis in Bangladesh. Trop Geogr Med. 1994;46(1):40-2. PMID 8165738
- [Background] Huilan S, Zhen LG, Mathan MM, Mathew MM, Olarte J, Espejo R, Khin Maung U, Ghafoor MA, Khan MA, Sami Z, et al. Etiology of acute diarrhoea among children in developing countries: a multicentre study in five countries. Bull World Health Organ. 1991;69(5):549-55. PMID 1659953
- [Background] Struelens MJ, Patte D, Kabir I, Salam A, Nath SK, Butler T. Shigella septicemia: prevalence, presentation, risk factors, and outcome. J Infect Dis. 1985 Oct;152(4):784-90. doi: 10.1093/infdis/152.4.784. PMID 4045231
- [Result] Passwell JH, Ashkenazi S, Banet-Levi Y, Ramon-Saraf R, Farzam N, Lerner-Geva L, Even-Nir H, Yerushalmi B, Chu C, Shiloach J, Robbins JB, Schneerson R; Israeli Shigella Study Group. Age-related efficacy of Shigella O-specific polysaccharide conjugates in 1-4-year-old Israeli children. Vaccine. 2010 Mar 2;28(10):2231-2235. doi: 10.1016/j.vaccine.2009.12.050. Epub 2010 Jan 5. PMID 20056180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: May 1, 2003 to January 31 3006. Surveillance period: May 1, 2003 to January 31 2008. Children were recruited from day care centers and health clinics in Israel
Groups:
- S. Sonnei Conjugate Vaccine: Shigella sonnei O-specific polysaccharide covalently bound to recombinant exoprotein A of Pseudomonas aeruginosa, administered in 2 injections of 0.5 mL containing 25 mcg of saccharide, 6 weeks apart
- S. Flexneri 2a Conjugate Vaccine: Shigella flexneri 2a O-specific polysaccharide covalently bound to recombinant exoprotein A of Pseudomonas aeruginosa, administered in 2 injections of 0.5 mL containing 25 mcg of saccharide, 6 weeks apart
Period: Overall Study
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine
Started | 1434 | 1365
Completed | 1392 | 1319
Not Completed | 42 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine | Total
Number analyzed (Participants) | 1434 | 1365 | 2799
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1434 | 1365 | 2799
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702 | 642 | 1344
  Male | 732 | 723 | 1455
Region of Enrollment [Number; unit: participants]
  Israel | 1434 | 1365 | 2799

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with events per vaccine type and dose occuring in >=5% of participants
Time Frame: Monitored for 7 days per participant following each injection for initial group of 500, 2 days for extended study of up to 5500 additional children
Measure: Number; unit: participants
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine
Number analyzed (Participants) | 1434 | 1365
participants
  local pain, dose 1 | 82 | 61
  local pain, dose 2 | 79 | 64
  fever, dose 1 | 56 | 72
  fever, dose 2 | 36 | 51

2. Secondary Outcome: Geometric Mean Immunoglobulin G (IgG) Anti-Lipopolysaccharide (LPS) Levels
Description: Age-related homologous IgG anti-LPS levels
Time Frame: Injections were administered 6 weeks apart and IgG anti-LPS levels determined >2 weeks after second vaccine dose. Each of the 15 sites also took a sample/week randomly chosen, for 2 years of follow up and blood samples from patients with disease
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine
Number analyzed (Participants) | 1434 | 1365
ELISA units
  Age 1-2 years | 1.40 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died. | 18.98 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died.
  Age >2-3 years | 3.71 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died. | 26.96 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died.
  Age >3-4 years | 6.38 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died. | 43.86 [NA to NA] — No measure of dispersion was calculated. The medically responsible investigator in Israel died.

3. Secondary Outcome: Percentage of Efficacy
Description: Percent efficacy is defined as ((disease rate of controls minus disease rate of vaccinees) divided by disease rate of controls) times 100
Time Frame: During 2 years post vaccination
Measure: Mean (95% Confidence Interval); unit: Percent efficacy
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine
Number analyzed (Participants) | 1434 | 1365
Percent efficacy
  Participants aged 1-2 years | 3.8 [-101.1 to 46.5] | -8.4 [-434.5 to 78.0]
  Participants aged >2-3 years | 35.5 [-56.4 to 73.4] | 22.5 [-244.4 to 82.6]
  Participants aged >3-4 years | 71.1 [-4.43 to 92.0] | -3.6 [-1550 to 93.5]

ADVERSE EVENTS:
Time Frame: Local and systemic reactions were sought at 30 minutes, 6, 24 and 48 hours after vaccination by a structured questionnaire.
Arm/Group | S. Sonnei Conjugate Vaccine | S. Flexneri 2a Conjugate Vaccine
Serious Adverse Events (participants affected / at risk) | 0/1434 | 0/1365
Other Adverse Events (participants affected / at risk) | 217/1434 | 197/1365
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S. Sonnei Conjugate Vaccine (N=1434) | S. Flexneri 2a Conjugate Vaccine (N=1365)
local pain, dose 1 (Musculoskeletal and connective tissue disorders) | 82 (82) | 61 (61)
local pain, dose 2 (Musculoskeletal and connective tissue disorders) | 79 (79) | 64 (64)
fever, dose 1 (Investigations) | 56 (56) | 72 (72)
fever, dose 2 (General disorders) | 36 (36) | 72 (72)

LIMITATIONS AND CAVEATS:
No efficacy could be assessed after 2nd injection of S. sonnei conjugate due to the small number of positive isolates at that time. There were too few cases of S. flexneri 2a infection for evaluation of vaccine B efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No